CLINICAL TRIAL: NCT00558025
Title: A Double-blind, Double-dummy, Randomized, Parallel Groups Study to Assess the Efficacy, Safety and Tolerability of Switching Patients With Early Parkinson's Disease (PD) From Pramipexole IR to Pramipexole ER or Pramipexole IR
Brief Title: Overnight Switch Trial From Pramipexole IR to Pramipexole ER in Patients With Early Parkinson Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.636; Eudract 2007-003353-90
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pramipexole Extended Release (ER) (Experimental): Pramipexole Extended Release (ER) once daily
  Interventions: Drug: Pramipexole Extended Release
- Pramipexole Immediate Release (IR) (Experimental): Pramipexole Immediate Release (IR) once daily
  Interventions: Drug: Pramipexole Immediate Release

INTERVENTIONS:
Drug: Pramipexole Extended Release
  Arms: Pramipexole Extended Release (ER)
Drug: Pramipexole Immediate Release
  Arms: Pramipexole Immediate Release (IR)

SUMMARY:
The objectives of this trial conducted in early Parkinson's disease (PD) patients are:

* To assess if patients with early Parkinson's disease (PD) can be successfully switched (overnight switching) from Pramipexole (PPX) Immediate Release (IR) to Pramipexole Extended Release (ER). A successful switch at a specific visit is defined as no worsening of the Unified Parkinsons Disease Rating Scale (UPDRS) parts II+III score by more than 15% from baseline and no drug-related adverse events leading to withdrawal;
* To establish if this successful switch can be obtained with or without dose-adaptation;
* To provide information about the conversion ratio (mg:mg) from Pramipexole IR to Pramipexole ER.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with idiopathic Parkinson's disease (PD) confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity.
2. Parkinson's disease diagnosed within 5 years.
3. Patients 30 years of age or older at the time of diagnosis.
4. Modified Hoehn and Yahr stage of 1 to 3.
5. Patients receiving pramipexole IR for at least three months prior to baseline visit (randomization visit, V2).
6. Pramipexole dose should be optimized (according investigator¿s judgement), greater or equal to 1.5 mg/day, stable and equally divided 3 times per day, for a least 4 weeks prior to baseline visit (V2).
7. Patients willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
8. Signed informed consent obtained before any study procedures are carried out in accordance with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines and local legislation).

Exclusion Criteria:

1. Motor complications under levodopa therapy at V1.
2. Atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases.
3. Dementia, as defined by a Mini-Mental State Exam score < 24 at V1
4. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria
5. History of psychosis, except history of drug induced hallucinations
6. Clinically significant electrocardiogram (ECG) abnormalities at V1.
7. Clinically significant hypotension either at screening visit or at baseline visit.
8. Malignant melanoma or history of previously treated malignant melanoma.
9. Any other clinically significant disease
10. Pregnancy or breast-feeding.
11. Sexually active female of childbearing potential
12. Serum levels of Aspartate Aminotransferase (Serum Glutamic Oxaloacetic Transaminase) (AST (SGOT)), Alanine Aminotransferase (Serum Glutamate Pyruvate Transaminase) (ALT (SGPT)), alkaline phosphatases or bilirubin > 2 Upper Limit of Normal (ULN) (on screening lab test).
13. Patients with a creatinine clearance < 50 mL/min
14. Any dopamine agonist (except pramipexole IR) within three months prior to baseline visit.
15. History of discontinuation of treatment with pramipexole IR
16. Previous treatment with pramipexole ER.
17. Any medication (including intra-muscular formulations) with central dopaminergic antagonist activity within 4 weeks prior to the baseline visit (i.e. typical neuroleptics, atypical antipsychotics, reserpine, methyldopa, centrally-active antiemetics, etc).
18. Any of the following drugs within 4 weeks prior to the baseline visit: methylphenidate, cinnarizine, amphetamines.
19. Flunarizine within 3 months prior to baseline visit.
20. Known hypersensitivity to Pramipexole or its excipients.
21. Drug abuse (including alcohol), according to Investigator¿s judgement, within 2 years prior to screening.
22. Participation in other investigational drug studies or use of other investigational drugs within 4 weeks or five times the half-life of the investigational drug (whichever is longer) prior to baseline visit.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- France (22):
  - 248.636.3303A Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.636.3303B Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.636.3303C Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.636.3307C Boehringer Ingelheim Investigational Site, Bron
  - 248.636.3309B Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 248.636.3305A Boehringer Ingelheim Investigational Site, Créteil
  - 248.636.3305B Boehringer Ingelheim Investigational Site, Créteil
  - 248.636.3313A Boehringer Ingelheim Investigational Site, Dijon
  - 248.636.3304A Boehringer Ingelheim Investigational Site, Évreux
  - 248.636.3308B Boehringer Ingelheim Investigational Site, Lille
  - 248.636.3308C Boehringer Ingelheim Investigational Site, Lille
  - 248.636.3308D Boehringer Ingelheim Investigational Site, Lille
  - 248.636.3308E Boehringer Ingelheim Investigational Site, Lille
  - 248.636.3302A Boehringer Ingelheim Investigational Site, Marseille
  - 248.636.3302B Boehringer Ingelheim Investigational Site, Marseille
  - 248.636.3306B Boehringer Ingelheim Investigational Site, Montpellier
  - 248.636.3312A Boehringer Ingelheim Investigational Site, Rouen
  - 248.636.3312B Boehringer Ingelheim Investigational Site, Rouen
  - 248.636.3311A Boehringer Ingelheim Investigational Site, Strasbourg
  - 248.636.3301A Boehringer Ingelheim Investigational Site, Toulouse
  - 248.636.3301B Boehringer Ingelheim Investigational Site, Toulouse
  - 248.636.3301D Boehringer Ingelheim Investigational Site, Toulouse
- Germany (8):
  - 248.636.49006 Boehringer Ingelheim Investigational Site, Achim Bei Bremen
  - 248.636.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 248.636.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 248.636.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 248.636.49002 Boehringer Ingelheim Investigational Site, Gera
  - 248.636.49001 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 248.636.49003 Boehringer Ingelheim Investigational Site, Steglitz
  - 248.636.49005 Boehringer Ingelheim Investigational Site, Unterhaching
- Netherlands (6):
  - 248.636.31005 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 248.636.31002 Boehringer Ingelheim Investigational Site, Geldrop
  - 248.636.31003 Boehringer Ingelheim Investigational Site, Helmond
  - 248.636.31006 Boehringer Ingelheim Investigational Site, Maastricht
  - 248.636.31004 Boehringer Ingelheim Investigational Site, Nijmegen
  - 248.636.31001 Boehringer Ingelheim Investigational Site, Sittard

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole Extended Release (ER): 0.375mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, 4.5mg, q.d. (Quaque die, once per day), per os
- Pramipexole Immediate Release (IR): 0.125 mg, 0.25 mg, 0.5 mg, 0.75 mg, 1.0 mg, 1.25 mg, 1.5 mg, t.i.d (Tres in die, three times daily), per os
Period: Overall Study
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Started | 104 | 52
Completed | 100 | 49
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pramipexole Extended Release (ER): 0.375mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, 4.5mg, q.d (Quaque die, once per day), per os
- Total: Total of all reporting groups
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR) | Total
Number analyzed (Participants) | 104 | 52 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (8.8) | 63.5 (9.7) | 63.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 21 | 68
  Male | 57 | 31 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Successfully Switched From Pramipexole Immediate Release (IR) to Pramipexole ER After a Possible Dose Adaptation, Full Analysis Set (FAS), Last Observation Carried Forward (LOCF)
Description: A successful switch was defined by no change of the Unified Parkinson's Disease Rating Scale (UPDRS) II+III by more than 15% from baseline to week 9, UPDRS II+III score ranging from 0 (no impairment) to 160 (worst impairment)
Time Frame: from baseline to week 9
Population: Full Analysis Set (FAS), all randomized patients that received treatment and had baseline and post baseline measurements for the primary endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
Percentage of participants
  Successfully switched | 84.5 | 94.2
  Not successfully switched | 15.5 | 5.8

2. Secondary Outcome: Percentage of Patients Who Successfully Switched From Pramipexole IR to Pramipexole ER With no Dose Adaptation, FAS (LOCF)
Description: A successful switch was defined by no change of the UPDRS II+III by more than 15% from baseline to week 4, UPDRS II+III score ranging from 0 (no impairment) to 160 (worst impairment).
Time Frame: from baseline to week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
Percentage of participants
  Successfully switched | 81.6 | 92.3
  Not successfully switched | 18.4 | 7.7
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Successfully switched patients; Test type: Non-Inferiority or Equivalence — Non-inferiority margin: -15 %, power: 80%; Wilson score interval; Risk Difference (RD) = -10.75, 95% CI [-20.51 to 1.48]
Statistical Analysis 2: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.0803, Cochran-Mantel-Haenszel; test with stratification by country

3. Secondary Outcome: Change From Baseline in UPDRS Part II+III Total Score at Week 9, FAS (LOCF)
Description: Unified Parkinson's Disease Rating Scale part II+III total score on FAS, Week 9 - baseline, UPDRS II+III score ranging from 0 (no impairment) to 160 (worst impairment)
Time Frame: Baseline and week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
Score on scale | -1.6 (0.5) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.2061, ANCOVA; ANCOVA with factors of treatment, country and baseline as covariate; Mean Difference (Final Values) = -1.1, 95% CI [-2.8 to 0.6]

4. Secondary Outcome: Change From Baseline in UPDRS Part II Total Score at Week 9, FAS (LOCF)
Description: Unified Parkinson's Disease Rating Scale part II total score on FAS, Week 9 - baseline, UPDRS II score ranging from 0 (no impairment) to 52 (worst impairment)
Time Frame: Baseline and week 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on Scale
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
Score on Scale | -0.3 (0.2) | -0.1 (0.3)
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.4694, ANCOVA; ANCOVA with factors of treatment, country and baseline as covariate; Mean Difference (Final Values) = -0.2, 95% CI [-0.8 to 0.4]

5. Secondary Outcome: Change From Baseline in UPDRS Part III Total Score at Week 9, FAS (LOCF)
Description: Unified Parkinson's Disease Rating Scale part III total score on FAS, week 9 - baseline, UPDRS II+III score ranging from 0 (no impairment) to 108 (worst impairment)
Time Frame: Baseline and week 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
Score on Scale | -1.2 (0.4) | -0.3 (0.6)
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.1804, ANCOVA; ANCOVA with factors of treatment, country and baseline as covariate; Mean Difference (Final Values) = -0.9, 95% CI [-2.3 to 0.4]

6. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I), FAS (LOCF)
Description: Clinical Global Impression - Improvement on FAS, CGI-I was rated from 1: very much improved, to 7: very much worse, CGI-I responder are defined as being rated as 'unchanged', 'minimally improved', 'much improved', or 'very much improved', CGI-I non-responder are defined as being rated 'minimally worse', 'much worse' or 'very much worse'
Time Frame: Week 9
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
participants
  CGI-I responder | 90 | 41
  CGI-I non-responder | 13 | 11
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.1623, Cochran-Mantel-Haenszel; test with stratification by country

7. Secondary Outcome: Patient Global Impression - Improvement (PGI-I), FAS (LOCF)
Description: Patient Global Impression - Improvement on FAS, PGI-I was rated from 1: very much better, to 7: very much worse, PGI-I responder are defined as being rated as 'unchanged', 'minimally better', 'much better', or 'very much better', PGI-I non-responder are defined as being rated as 'minimally worse', 'much worse', or 'very much worse'
Time Frame: Week 9
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
participants
  PGI-I responder (unchanged to very much better) | 84 | 37
  PGI-I non-responder | 19 | 15
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.1299, Cochran-Mantel-Haenszel; test with stratification by country

8. Secondary Outcome: Pramipexole Dose Adaptation, FAS (LOCF)
Description: Patients with increase in daily Pramipexole dose on FAS
Time Frame: Week 9
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 103 | 52
participants
  Daily dose increased | 17 | 7
  Daily dose not increased | 86 | 45
Statistical Analysis 1: Comparison: Pramipexole Extended Release (ER) vs Pramipexole Immediate Release (IR); Test type: Superiority or Other; p = 0.6190, Cochran-Mantel-Haenszel; test with stratification by country

9. Secondary Outcome: Final Pramipexole Dose (mg) After 9 Weeks, Treated Set
Description: The mean final daily Pramipexole dose is displayed
Time Frame: Week 9
Population: Treated Set (TS) includes all patients randomized and who received treatment
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Number analyzed (Participants) | 104 | 52
mg | 2.75 (0.95) | 2.83 (0.86)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Pramipexole Extended Release (ER) | Pramipexole Immediate Release (IR)
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/52
Other Adverse Events (participants affected / at risk) | 0/104 | 0/52

LIMITATIONS AND CAVEATS:
There were no serious adverse events in the trial and no non-serious adverse events with an incidence >5%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.